CLINICAL TRIAL: NCT00134238
Title: Phase 3 Multi-Center, Double-Blind, Randomized, Parallel Group, Carotid B-mode Ultrasound Evaluation of the Anti-Atherosclerotic Efficacy, Safety, and Tolerability of Fixed Combination CP-529,414/Atorvastatin, Administered Orally, Once Daily (QD) for 24 Months, Compared With Atorvastatin Alone, in Subjects With Mixed Hyperlipidemia
Brief Title: Carotid B-mode Ultrasound Study to Compare Anti-Atherosclerotic Effect of Torcetrapib/Atorvastatin to Atorvastatin.
Acronym: RADIANCE 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091004
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To look at ultrasound images taken in the carotid arteries and to look at various lipids in the blood of people with mixed hyperlipidemia

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mixed hyperlipidemia
* At least 18 years of age

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid (high doses)
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluationof response, or render unlikely that the subject would complete the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in intima media thickness as measured by carotid ultrasound

SECONDARY OUTCOMES:
Changes in levels of lipids and other biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (40):
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Alhambra, California
  - Pfizer Investigational Site, Encinitas, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Palm Bay, Florida
  - Pfizer Investigational Site, Sebastian, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Cambridge, Massachusetts
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Concord, New Hampshire
  - Pfizer Investigational Site, Bronxville, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Mount Vernon, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Bothell, Washington
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Seattle, Washington
- Canada (5):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, Prague, Czechia
- Pfizer Investigational Site, Kuopio, Finland
- Pfizer Investigational Site, Paris, France
- Netherlands (3):
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Utrecht

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- [Derived] Tajik P, Meijer R, Duivenvoorden R, Peters SA, Kastelein JJ, Visseren FJ, Crouse JR 3rd, Palmer MK, Raichlen JS, Grobbee DE, Bots ML. Asymmetrical distribution of atherosclerosis in the carotid artery: identical patterns across age, race, and gender. Eur J Prev Cardiol. 2012 Aug;19(4):687-97. doi: 10.1177/1741826711410821. Epub 2011 May 25. PMID 21613319
- [Derived] Vergeer M, Bots ML, van Leuven SI, Basart DC, Sijbrands EJ, Evans GW, Grobbee DE, Visseren FL, Stalenhoef AF, Stroes ES, Kastelein JJ. Cholesteryl ester transfer protein inhibitor torcetrapib and off-target toxicity: a pooled analysis of the rating atherosclerotic disease change by imaging with a new CETP inhibitor (RADIANCE) trials. Circulation. 2008 Dec 9;118(24):2515-22. doi: 10.1161/CIRCULATIONAHA.108.772665. Epub 2008 Nov 24. PMID 19029469
- [Derived] Bots ML, Visseren FL, Evans GW, Riley WA, Revkin JH, Tegeler CH, Shear CL, Duggan WT, Vicari RM, Grobbee DE, Kastelein JJ; RADIANCE 2 Investigators. Torcetrapib and carotid intima-media thickness in mixed dyslipidaemia (RADIANCE 2 study): a randomised, double-blind trial. Lancet. 2007 Jul 14;370(9582):153-160. doi: 10.1016/S0140-6736(07)61088-5. PMID 17630038
- [Derived] Kastelein JJ, van Leuven SI, Evans GW, Riley WA, Revkin JH, Shear CL, Bots ML; RADIANCE 1 and 2 Study Investigators. Designs of RADIANCE 1 and 2: carotid ultrasound studies comparing the effects of torcetrapib/atorvastatin with atorvastatin alone on atherosclerosis. Curr Med Res Opin. 2007 Apr;23(4):885-94. doi: 10.1185/030079907x182121. PMID 17407645